CLINICAL TRIAL: NCT06033729
Title: Remifentanil Target Controlled Infusion Versus Standard of Care for Conscious Sedation During US-guided Transbronchial Needle Aspiration (EBUS-TBNA): a Randomized, Prospective, Control Study
Brief Title: Remifentanil Target Controlled Infusion Versus Standard of Care for Conscious Sedation During EBUS-TBNA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scarlata, Simone, M.D. (Other)
Responsible Party: Principal Investigator, Simone Scarlata, Associate Professor in Internal Medicine, Scarlata, Simone, M.D.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CBM 20-12
Record Dates: First submitted 2023-08-21; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Lung Cancer; Lung; Node; Sedation Complication; Endoscopy
Keywords: endobronchial ultrasound; mediastinal staging of lung cancer; sedation in endoscopic procedures
MeSH Terms: conditions — Lung Neoplasms | interventions — Midazolam; Fentanyl; Propofol

STUDY DESIGN:
Intervention Model Description: Informed consent was obtained from each patient or legally authorized representative prior to enrollment in this study.
  After obtaining a signed informed consent the patient was randomly allocated 1:1 to the group "REMIFENTANIL TCI" or "STANDARD". A research randomizer software was used for randomization (iRANDOMIZER-SHMOOPI LLC-version 2.5).
Who Masked: Participant, Outcomes Assessor
Masking Description: The bronchoscopist, the patient and the research assistant administrating the questionnaires were blinded to the assigned group. It was not possible to blind anesthesiologists involved in the patient's care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 "REMIFENTANIL TCI" (Experimental Group) (Experimental): the patients performed the EBUS-TBNA procedure under conscious sedation with infusion of Remifentanil TCI with a target between 3 and 6 ng/ml;
  Interventions: Drug: Remifentanil TCI
- Group 2 "STANDARD" (Control Group) (Active Comparator): the patients performed the EBUS-TBNA procedure in conscious sedation with the association of midazolam and/or fentanyl and/or propofol in refracted boluses based on clinical needs (agitation, unsatisfactory level of sedation or not collaborative patient) and according to the anesthesiologist's clinical judgement.
  Interventions: Drug: Midazolam injection; Drug: Fentanyl; Drug: Propofol

INTERVENTIONS:
Drug: Remifentanil TCI — REMI-TCI administration begun 5 minutes before the procedure, starting from an initial target at the effect site of 1 ng/ml and gradually increasing by 0.5 ng/ml until reaching an adequate level of sedation (Ramsey score between 2-3).
  Other Names: REMI - target control infusion
  Arms: Group 1 "REMIFENTANIL TCI" (Experimental Group)
Drug: Midazolam injection — Bolus administration of midazolam (1-2 mg)and/or until a Ramsey score 2-3 was reached
  Other Names: Bolus administration of midazolam
  Arms: Group 2 "STANDARD" (Control Group)
Drug: Fentanyl — Bolus adminitration of fentanyl (50-100 mcg) until a Ramsey score 2-3 was reached
  Other Names: Bolus administration of Fentanyl
  Arms: Group 2 "STANDARD" (Control Group)
Drug: Propofol — Bolus adminitration of propofol until a Ramsey score 2-3 was reached
  Other Names: Bolus administration of Propofol
  Arms: Group 2 "STANDARD" (Control Group)

SUMMARY:
Background: endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA) is a minimally invasive procedure for diagnosing and staging mediastinal lymph node lesions in lung cancer. Adequate sedation is crucial for patient comfort and diagnostic accuracy. Different sedation modalities, including moderate sedation/conscious sedation, deep sedation, and general anesthesia, are utilized. This study aims to evaluate patient comfort and satisfaction levels of healthcare providers (bronchoscopists and anesthesiologists) when administering remifentanil through Target Controlled Infusion (TCI) for conscious sedation during EBUS-TBNA. A prospective randomized study design compares this approach to the standard sedation protocol involving midazolam, fentanyl, and/or propofol.

Methods: this study will enroll 30 eligible patients randomly divided into two groups. Group 1, "REMIFENTANIL TCI", underwent EBUS-TBNA under conscious sedation with remifentanil TCI infusion targeting a concentration of 3-6 ng/ml. Group 2, "STANDARD", received conscious sedation with a combination of midazolam, fentanyl, and/or propofol administered in boluses based on clinical requirements. Complications, safety, and satisfaction levels of the operator, anesthesiologist, and patients will be evaluated.

DETAILED DESCRIPTION:
BACKGROUND Endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA) is a minimally invasive procedure that has gained major relevance in diagnosis lung cancer and staging of mediastinal lymph nodes (LN). Adequate sedation is an important part of the procedure since it improves patient's comfort and tolerance potentially positively affecting the diagnostic yield. It is also considered a standard of care for patients undergoing fiberoptic bronchoscopy unless specifically contraindicated.

The choice of the different level of sedation (from conscious to moderate to deep sedation) has always been challenging and, to date, no standardized practice exists. Deep sedation may be preferred in those cases where additional procedures such as placement of endobronchial stents, are required, or in order to make the procedure more suitable by limiting the patients motion. In remaining cases, conscious sedation allows to complain with the clinical demand without affecting respiratory and cardiovascular function, decreasing the cough reflex and maintaining sufficient swallowing capacity.

Not appropriate sedation can have serious complications, including respiratory depression or even arrest, hypoxia and/or hypercapnia, and cardiovascular and neurological side effects.

Commonly used drugs for sedation include propofol and a combination of benzodiazepines and opioids. However, achieving the ideal level of sedation can be challenging, since it may occasionally lead to over sedation, with detrimental effects. These risks are even greater if the patients present with lung disease, obesity, or heart disease. Conversely, under sedation can result in discomfort for the patient and challenging procedure it for the healthcare provider. Furthermore, benzodiazepines and medium-long-acting opioids continue their effect even after the procedure is finished, thus lasting the negative effects of these drugs over the time of the procedure.

In a recent case series, Scarlata and colleagues have provided a preliminary evidence of a TCI remifentanil protocol safety and effectiveness, providing an ideal and performant condition for bronchoscopists and a satisfactory comfort for patients.

Using a TCI continuous infusion protocol of Remifentanil can exploit the sedative, analgesic and antitussive capabilities of this short-acting opioid, achieving a level of conscious sedation that ensures an adequate level of comfort for the patient while at the same time decreases the incidence of side effects typical of deep sedation. The patient remains contactable and can respond and execute commands, such as breathing, swallowing, etc.

TCI is a method of continuous drug administration where the infusion of the drug is remotely controlled. There are different administration algorithms and there is the possibility to titrate the target concentration both at the effect site (CNS) and in the plasma.

There are numerous studies confirming the efficacy of remifentanil administered by TCI during intubation with an awake patient, and the advantages of the latter compared to other techniques, such as propofol infusion. One study determined the efficacy of infused remifentanil and propofol for bronchial endoscopy procedures, but did not use the TCI technique for infusion. There are no clinical studies assessing endoscopic transbronchial needle biopsy procedures with remifentanil infusion in TCI mode.

The aim of this study is therefore to conduct a prospective, randomized, controlled trial to evaluate the administration of remifentanil in TCI for conscious sedation during EBUS-TBNA procedures, the degree of patient and operator satisfaction and the relative advantages and disadvantages versus the of standard sedation protocol with midazolam and/or fentanyl and/or propofol.

METHODS This is a single center, randomized, investigator initiated clinical trial of 30 patients undergoing EBUS-TBNA for mediastinal staging of lung cancer. Patients were randomly assigned to one of two groups: Group 1 "REMIFENTANIL TCI" (Experimental Group): the patients performed the EBUS-TBNA procedure under conscious sedation with infusion of Remifentanil TCI with a target between 3 and 6 ng/ml; Group 2 "STANDARD" (Control Group): the patients performed the EBUS-TBNA procedure in conscious sedation with the association of midazolam and/or fentanyl and/or propofol in refracted boluses based on clinical needs (agitation, unsatisfactory level of sedation or not collaborative patient) and according to the anesthesiologist's clinical judgement.

After obtaining a signed informed consent the patient was randomly allocated 1:1 to the group "REMIFENTANIL TCI" or "STANDARD". A research randomizer software was used for randomization (iRANDOMIZER-SHMOOPI LLC-version 2.5). Both the bronchoscopist and the research assistant administrating the questionnaires were blinded to the assigned group. It was not possible to blind anesthesiologists involved in the patient's care.

The procedures used in this study adhere to the tenets of the Declaration of Helsinki.

Study treatment The ASA scale, the Mallampati score, the presence of OSAS were recorded prior of the procedure. Also, data about the underlying oncological disease, whether chemotherapy and/or radiotherapy was performed, and the indication for the EBUS-TBNA test (diagnostic, staging, re-staging, or both diagnostic and staging at the same moment) were collected.

The patient candidate for the endoscopic procedure underwent continuous monitoring of vital signs. ECG with precordial leads, continuous finger pulse oximetry, and noninvasive intermittent blood pressure measurements were monitored. Each patient was preoxygenated for about 5 minutes by administering O2 with nasal goggles at 3L/min or higher, if required.

Lidocaine was topically nebulized at the level of the mucous membranes of the oropharynx. Oxybuprocaine 4mg/ml was also nebulized at the level of the vocal cords via the eco-endoscope before passing the glottic plane in all patients.

Remifentanil group conscious sedation protocol (intra venous remifentanil in TCI). Drug administration begun 5 minutes before the procedure. The achievement of the ideal target occurs starting from an initial target at the effect site of 1 ng/ml and gradually increasing the desired target on the pump by 0.5 ng/ml at a time, until reaching a target between 3 and 6 ng/ml and an adequate level of sedation (Ramsey Score between 2-3).

Desired target was achieved by automatic infusion pumps (Infusomat® Space® Large Volume Pump, Braun medical inc) If, despite the maximum target, a satisfactory level of sedation was not reached, repeated boluses of propofol were given as clinically needed and the case considered as protocol failure.

Patients in the STANDARD Group performed the EBUS-TBNA with bolus administration of midazolam and/or fentanyl and/or propofol. Shortly before the start of the procedure they received 1-2 mg bolus midazolam and/or 50-100 range bolus fentanyl until they reach the level of sedation (Ramsey Score 2-3). In addition, repeated boluses of propofol could have been given according to clinical needs (state of agitation of the patient, requests from the operator due to difficulties in carrying out the procedure).

Data were collected about the procedure performed, any changes in vital signs that occurred during the procedure and the depth of sedation.

Anesthesiologist, bronchoscopist and patient's satisfaction tools At the end of the procedure, the patient was given a satisfaction questionnaire to evaluate the degree of satisfaction. The 0-5 Likert numerical scale was used to evaluate the symptoms onset of cough (0 none-5 very much), sore throat (0-5), chest pain (0-5), shortness of breath (0 eupnoea- 5 worsening dyspnea), presence of memories (0 none - 5 vivid memories), and perioperative comfort (0 none - 5 excellent). The operator who performed the procedure and the sedation were also subjected to a satisfaction questionnaire which assessed the overall satisfaction (1 much worse than usual - 5 much better than usual).

Statistical Analysis The analysis was performed on an intention to treat basis, regardless of actual compliance with the intended intervention.

A two-tailed p value equal or less than 0.05 was considered as statistically significant. All tests, except for the primary outcome, were considered merely exploratory. When individual items were missing from a scale, the percent of missing values and, if more than 10% was calculated, the scale score was considered missing and therefore made unavailable for analysis. All the analyses were conducted using STATA (StataCorp. 2021. Stata Statistical Software: Release 17. College Station, TX: StataCorp LLC.).

Outcome analysis Primary and secondary endpoints will be compared between the two groups of treatment by means of Student's t-test (or the Mann-Whitney U test, if necessary) for continuous quantitative variables and by means of the χ2 test (or Fisher's exact test ) for qualitative variables.

Sample size determination Our previously published case series showed that the overall satisfaction rate for both the patient and the bronchoscopist were very high in the remifentanil TCI group (mean Likert score above 4/5 against a mean value ranging from 2 to 3 in the standard group as available in the literature). Enrolling 30 patients (fifteen for each group) would have provided with 80% power at an alpha level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18-80 years,
* clinical fit to undergo the planned procedure, according to the American Society of Anesthesiologists physical status classification.

Exclusion Criteria:

* current chronic opioid treatment,
* substance abuse or drug use;
* pregnancy,
* history of allergy to related medications;
* severe coagulation dysfunction;
* severe hepatic
* renal dysfunction;
* history of abnormal recovery from anesthesia;
* acute respiratory failure;
* inability or unwillingness to provide informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2023-01-17 (Actual)

PRIMARY OUTCOMES:
Patient, bronchoscopist and anesthesiologist's comfort and satisfaction to the procedure. | At patient's dismission from bronchoscopy suit
  the patient was given a satisfaction questionnaire to evaluate the degree of satisfaction. The 0-5 Likert numerical scale was used to evaluate the symptoms onset of cough (0 none-5 very much), sore throat (0-5), chest pain (0-5), shortness of breath (0 eupnoea- 5 worsening dyspnea), presence of memories (0 none - 5 vivid memories), and perioperative comfort (0 none - 5 excellent). The operator who performed the procedure and the sedation were also subjected to a satisfaction questionnaire which assessed the overall satisfaction (1 much worse than usual - 5 much better than usual).

SECONDARY OUTCOMES:
propofol boluses administered | During the procedure
  Number and dosage of any propofol boluses administered (both in the experimental group and in the control group)
Procedure time | During the procedure
  Total duration of the procedure (in minutes)
Level of sedation | During the procedure
  Level of sedation achieved (Ramsey score)
Over sedation | During the procedure
  Episodes of over-sedation (Ramsey score > 3)
Desaturation | Up to an hour from the end of the procedure
  Desaturation episodes
Hypotension | Up to an hour from the end of the procedure
  Episodes of hypotension (SBP <90 mmHg)
Bradycardia | Up to an hour from the end of the procedure
  Episodes of Bradycardia (HR<60)
Bradypnea or respiratory arrest | Up to an hour from the end of the procedure
  Episodes of bradypnea (RR<10)
Cough | Up to two hours from the end of the procedure
  Excessive cough (Unconfortable, unconstrained cough affecting patient's and operator comfort)
Airway support | Up to an hour from the and of the procedure
  Need for airway support
Sampled lymph nodes | During the procedure
  Number of lymph nodes sampled during the procedure.
Sampled lesions | During the procedure
  Number of masses sampled during the procedure.
Number of biopsies per limph node | During the procedure
  Number of biopsies per single lymph node needed to obtain a confident sample size according to a visual on-site evaluation.
Number of biopsies per mass | During the procedure
  Number of biopsies per single mass needed to obtain a confident sample size according to a visual on-site evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Università Campus Bio Medico, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wahidi MM, Jain P, Jantz M, Lee P, Mackensen GB, Barbour SY, Lamb C, Silvestri GA. American College of Chest Physicians consensus statement on the use of topical anesthesia, analgesia, and sedation during flexible bronchoscopy in adult patients. Chest. 2011 Nov;140(5):1342-1350. doi: 10.1378/chest.10-3361. PMID 22045879
- [Result] Aswanetmanee P, Limsuwat C, Kabach M, Alraiyes AH, Kheir F. The role of sedation in endobronchial ultrasound-guided transbronchial needle aspiration: Systematic review. Endosc Ultrasound. 2016 Sep-Oct;5(5):300-306. doi: 10.4103/2303-9027.191608. PMID 27803902
- [Result] Scarlata S, Costa F, Pascarella G, Strumia A, Antonelli Incalzi R, Agro FE. Remifentanil Target-Controlled Infusion for Conscious Sedation in Endobronchial Ultrasound-Guided Transbronchial Needle Aspiration (EBUS-TBNA): A Case Series. Clin Drug Investig. 2020 Oct;40(10):985-988. doi: 10.1007/s40261-020-00960-0. No abstract available. PMID 32767252